CLINICAL TRIAL: NCT05370963
Title: Dexmedetomidine or Hyalase : Which of Them Can Augment Lumbar Epidural Steroid Injection in Failed Back Surgery Patients. A Randomized Clinical Trial
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Minia University (Other)
Responsible Party: Principal Investigator, Mina Maher, Lecturer of anesthesia and ICU, Minia University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 278/5-2022
Record Dates: First submitted 2022-05-07; First posted 2022-05-12 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-06

CONDITIONS: Pain, Chronic
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- hyalase group (Active Comparator): Bupivacaine 5 mg (1 mL) + Triamcinolone 40 mg (1 mL) + Saline solution (2 mL) + Hyaluronidase 1,500 IU reconstituted in 1 mL distilled water (HYL)
  Interventions: Drug: Hylase versus dexmedtemodine
- dexmedtemodine group (Active Comparator): Bupivacaine 5 mg (1 mL) + Triamcinolone 40 mg (1 mL) + Saline solution (2 mL) + Dexmedetomidine 0.5 mic/kg
  Interventions: Drug: Hylase versus dexmedtemodine

INTERVENTIONS:
Drug: Hylase versus dexmedtemodine — fluroscopic guided lumber epidural injection

SUMMARY:
hyalase and dexmedtemodine are well known adjuvants given epidurally to alleviate chronic back pain. Use in failed back surgery is an up to date field to hasten analgesia and py off recurrence .

ELIGIBILITY:
Inclusion Criteria:

* Age group. 25-75ys old
* Both sex.
* persistent (at least 6 month) pain and or disability following laminectomy with or without sensory-motor neurological deficits or any form of urinary or bowel incontinence
* Patients suffering from persistent (> 6 months) back pain following laminectomy for spinal canal stenosis and/or discectomy for herniated nucleus pulposus documented by magnetic resonance imaging (MRI) were included for screening and enrollment.

Exclusion Criteria:

* Diabetic patients.
* Refusal to participate
* MRI with disc sequestration, concurrent sacro-ilitis, facet arthropathy .
* Coagulopathic patients
* Surgical induced discitis.

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2022-05-20 (Actual); Primary Completion 2023-05-30 (Actual); Study Completion 2023-06-01 (Actual)

PRIMARY OUTCOMES:
pain assesment | 6 months
  Visual analogue scale... 0= no pain .... 10= worst pain

SECONDARY OUTCOMES:
functional disability | 6 months
  Modified oswestry diability questionnaire. 0% to 20%: minimal disability:....21%-40%: moderate disability: 41%-60%: severe disability...61%-80%: crippled
acute complications | 6 hours
  number of patients with epidural hematoma

CONTACTS AND LOCATIONS:
Locations (1):
- Maher Maher, ALMinya, Egypt, Egypt